CLINICAL TRIAL: NCT00297960
Title: Influence of Treatment With Olanzapine or Ziprasidone on Transcapillary Glucose Transport in Human Skeletal Muscle
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: olanz/zipra; EUDRACT Nr.: 2004-002147-27
Record Dates: First submitted 2006-02-28; First posted 2006-03-01 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2005-10

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — ziprasidone; Olanzapine; Microdialysis

INTERVENTIONS:
Drug: ziprasidone or olanzapine
Procedure: hyperinsulinaemic euglycaemic clamp
Procedure: microdialysis (skeletal muscle)

SUMMARY:
Healthy volunteers will undergo euglycaemic hyperinsulinaemic clamp and microdialysis before and after administration of 10mg olanzapine or 80mg ziprasidone during 10 days.

DETAILED DESCRIPTION:
Background:

The efficacy of atypical antipsychotics, such as olanzapine, clozapine, risperidone, quetiapine and ziprasidone in treating a broad spectrum of symptoms in schizophrenia as well as their lower likelihood of extrapyramidal symptoms have led to an increased use of these substances. However there is an ongoing debate whether treatment with atypical antipsychotics is associated with a higher risk for metabolic abnormalities. The FDA stated in 2003 that all atypical antipsychotics increase the risk for glucose abnormalities. For olanzapine many, but not all studies report an increased risk for the development of metabolic abnormalities, such as glucose intolerance, insulin-resistance and consequentially NIDDM (Non-Insulin-Dependent-Diabetes Mellitus). Ziprasidone on the other hand seems to be associated with a more favorable metabolic safety profile.Glucose intolerance and insulin resistance being risk factors for the development of NIDDM and cardiovascular disease, the exact determination of putative effects of atypical antipsychotics on insulin sensitivity and resistance is of great need. An innovative technique, microdialysis, allows for the measurement of various analytes in the interstitial space, i.e. to assess insulin sensitivity directly at the responsible compartment, which is the human skeletal muscle. With the use of microdialysis it is possible to determine the arterial to interstitial gradient, a suitable marker for plasma glucose extraction of peripheral tissue, and thus detect insulin resistance directly at the site of insulin action.

Aim of the study:

To compare the effects of treatment with the atypical antipsychotics olanzapine and ziprasidone in steady-state conditions on the arterial to interstitial skeletal muscle gradient for glucose in human skeletal muscle during euglycaemic hyperinsulinaemic clamp conditions in male healthy volunteers.

Study design:

Open, randomized, mono-center study.

Materials and methods:

Healthy volunteers will undergo euglycaemic hyperinsulinaemic clamp and microdialysis before and after administration of 10mg olanzapine or 80mg ziprasidone during 10 days.

Study population:

15 healthy volunteers will participate in each arm of the study, summing up to a total of 30 participants.

Main outcome variable:

The arterial to interstitial skeletal muscle glucose gradient before and during euglycaemic hyperinsulinaemic clamp conditions, before and after administration of 10mg olanzapine or 80mg ziprasidone under steady-state conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-55
* Healthy male volunteers
* No history of drug or alcohol abuse
* No regular nicotine consumption at time of enrollment
* Physical activity at least twice a week
* Body mass Index between 19-24 kg/m2
* Normal laboratory values
* Normotension (blood pressure less than 140/90)
* No past or present history of psychiatric disorder
* No family history of diabetes or obesity
* Written informed consent

Exclusion Criteria:

* Use of medication within the last 14 days
* Consumption of alcohol within the last 5 days
* Family history of diabetes or obesity
* Past or present psychiatric disorder

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Siegfried Kasper, Prof. MD, Principal Investigator — Medical University Vienna, Department of General Psychiatry
Locations (1):
- Department of Clinical Pharmacology, Medical University Vienna, Vienna, Austria

REFERENCES:
- [Background] Newcomer JW, Haupt DW, Fucetola R, Melson AK, Schweiger JA, Cooper BP, Selke G. Abnormalities in glucose regulation during antipsychotic treatment of schizophrenia. Arch Gen Psychiatry. 2002 Apr;59(4):337-45. doi: 10.1001/archpsyc.59.4.337. PMID 11926934
- [Background] Rosdahl H, Lind L, Millgard J, Lithell H, Ungerstedt U, Henriksson J. Effect of physiological hyperinsulinemia on blood flow and interstitial glucose concentration in human skeletal muscle and adipose tissue studied by microdialysis. Diabetes. 1998 Aug;47(8):1296-301. doi: 10.2337/diab.47.8.1296. PMID 9703331
- [Background] Muller M, Holmang A, Andersson OK, Eichler HG, Lonnroth P. Measurement of interstitial muscle glucose and lactate concentrations during an oral glucose tolerance test. Am J Physiol. 1996 Dec;271(6 Pt 1):E1003-7. doi: 10.1152/ajpendo.1996.271.6.E1003. PMID 8997218